CLINICAL TRIAL: NCT05411250
Title: Early Diagnosis of Therapy-associated Cardiotoxicity Basing on PET/CT in Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Principal INvestigaor, Peking University Cancer Hospital & Institute
Other Study IDs: XW-Heart-002
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Positron-Emission Tomography
Keywords: cardiotoxicity; early
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the value of 18F-fluorodeoxyglucose (FDG) PET/CT imaging in early diagnosis of treatment-related cardiotoxicity (TACT) of lymphoma using visual method and semi-quantitative method.

DETAILED DESCRIPTION:
First of all, the cardiac 18F-FDG uptake in patients with lymphoma will be observed by visual method: according to the uptake site, it will be divided into left ventricular uptake and biventricular uptake, and according to the degree of uptake, it will be divided into equal uptake (myocardial uptake is lower than cardiac blood pool uptake), moderate uptake (myocardial uptake is between cardiac blood pool uptake and liver uptake) and high uptake (myocardial uptake is higher than liver uptake). According to the uptake pattern, it can be divided into diffuse and segmental uptake.Then,using the region of interest method to mesure the value of myocardial uptake of 18F-FDG.The difference value of heart's SUVmax (Δ SUVmax- heart) and% Δ SUVmax- heart before and after chemotherapy or immunotherapy will be calculated. And SUVmax- heart / SUVmax- mediastinum ratio, SUVmax- heart / SUVmax- liver ratio and SUVmax- heart / SUVmax- background ratio (left gluteal muscle) after treatment. Taking the abnormality of ECG (early TACT) as the end point.

ELIGIBILITY:
Inclusion Criteria:

1. No previous history of heart disease.
2. normal echocardiography, ECG and laboratory tests (creatine kinase, myoglobin, troponin, brain natriuretic peptide) before treatment.

3.18F-FDG PET/CT examination before and after treatment

-

Exclusion Criteria:

1.receiving radiotherapy and chemotherapy at the same time. 2.previous chest radiotherapy. 3. with severe hepatic or renal dysfunction.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumor after chemotherapy or immunotherapy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 150 days
  the standardized uptake value

SECONDARY OUTCOMES:
SUVR | 150 days
  the ratio of the standardized uptake value for the heart to the normal tissue such as hepatic blood poor and gluteus

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, PhD, Study Director — Peking cancer hospital

IPD SHARING:
Plan to Share IPD: No